CLINICAL TRIAL: NCT05080621
Title: A Phase 1b/2, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Ripretinib in Combination With Binimetinib in Patients With Gastrointestinal Stromal Tumor (GIST)
Brief Title: Ripretinib in Combination With Binimetinib in Patients With Gastrointestinal Stromal Tumor (GIST)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue this study due to a corporate restructuring intended to prioritize clinical development of select programs. No patients enrolled in this study and no patients received investigational product.
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2618-01-008
Record Dates: First submitted 2021-09-20; First posted 2021-10-18 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): Escalation Phase: Increasing doses of ripretinib in combination with increase doses of binimetinib in patients with advanced GIST who have progressed on at least imatinib or are intolerant to imatinib and are ripretinib naïve in repeated 28-day cycles.
  Participants may remain on treatment until disease progression, unacceptable toxicity, or withdrawal of consent
  Interventions: Drug: Ripretinib; Drug: binimetinib
- Expansion (Experimental): Ripretinib in combination with binimetinib at the recommended Phase 2 dose (RP2D) in patients with advanced GIST who have progressed on imatinib or are intolerant to imatinib and are naïve.
  Participants may remain on treatment until disease progression, unacceptable toxicity, or withdrawal of consent
  Interventions: Drug: Ripretinib; Drug: binimetinib

INTERVENTIONS:
Drug: Ripretinib — 50 mg tablets
  Other Names: DCC-2618, QINLOCK
Drug: binimetinib — 15 mg tablets
  Other Names: Mektovi

SUMMARY:
Multicenter, open-label Phase 1b/2 study of ripretinib in combination with binimetinib in patients with gastrointestinal stromal tumor (GIST). There will be 2 distinct parts in this study: Dose Escalation (Phase 1) and Expansion (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age with advanced GIST (unresectable or metastatic).
2. Must have at least progressed on imatinib or have documented intolerance to imatinib.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
4. Patients must have a histologic diagnosis of GIST.
5. If a female of childbearing potential, must have a negative pregnancy test.
6. Adequate organ function and bone marrow function

Exclusion Criteria:

1. Received prior anticancer therapy within 14 days or 5× the half-life whichever is longer) prior to the first dose.
2. Ongoing or prior participation in the DCC-2618-03-002 study.
3. Prior therapy with ripretinib.
4. Prior therapy with MEK inhibitor.
5. History of certain ocular disorders.
6. History of clinically significant hepatobiliary disease.
7. Known active central nervous system metastases.
8. History or presence of clinically relevant cardiovascular abnormalities.
9. Systemic arterial or venous thrombotic or embolic events within 6 months of first dose.
10. History of acute or chronic pancreatitis
11. History of chronic inflammatory bowel disease or Crohn's disease requiring intervention within 12 months of first dose.
12. Gastrointestinal abnormalities including but not limited to:

    * inability to take oral medication,
    * malabsorption syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety/tolerability of oral ripretinib in combination with binimetinib: incidence of adverse events | Approximately 12 months
  Adverse events [TEAEs, SAEs, AESIs], dose reduction, dose interruption, or discontinuation, vital signs (heart rate [beats/min], and changes in laboratory parameters (chemistry, hematology, urinalysis, coagulation).
Determination of the Maximum Tolerated Dose and the Recommended Phase 2 Dose | Approximately 12 months
Expansion Phase Only: Evaluate the objective response rate (ORR) of ripretinib in combination with binimetinib by modified RECIST | Approximately 36 months
  Measure ORR

SECONDARY OUTCOMES:
Determine the time to maximum observed concentration (tmax) profile of oral ripretinib in combination with binimetinib | Cycle 1 Day 1, and Cycle 1 Day15 (pre-dose and at multiple time points [up to 8 hours] post-dose). Each cycle is 28 days
  Measure Tmax
Determine the maximum observed concentration (Cmax) profile of oral ripretinib in combination with binimetinib | Cycle 1 Day 1, and Cycle 1 Day15 (pre-dose and at multiple time points [up to 8 hours] post-dose). Each cycle is 28 days
  Measure Cmax
Determine the minimum observed concentration (Cmin) profile of oral ripretinib in combination with binimetinib | Cycle 1 Day 1, and Cycle 1 Day15 (pre-dose and at multiple time points [up to 8 hours] post-dose). Each cycle is 28 days
  Measure Cmin
Determine the area under the concentration-time curve (AUC) profile of oral ripretinib in combination with binimetinib | Cycle 1 Day 1, and Cycle 1 Day15 (pre-dose and at multiple time points [up to 8 hours] post-dose). Each cycle is 28 days
  Measure AUC
Evaluate the objective response rate (ORR) of ripretinib in combination with binimetinib by modified RECIST (escalation phase only) and Choi criteria (escalation and expansion phases) | Approximately 36 months
  Measure ORR
Evaluate the progression-free survival (PFS) of ripretinib in combination with binimetinib | Approximately 36 months
  Measure PFS
Evaluate the overall survival (OS) of ripretinib in combination with binimetinib | Approximately 36 months
  Measure OS
Evaluate the duration of response (DOR) of ripretinib in combination with binimetinib | Approximately 36 months
  Measure DOR
Evaluate the clinical benefit rate (CBR) of ripretinib in combination with binimetinib | Approximately 36 months
  Measure CBR
Evaluate the time to response (TTR) of ripretinib in combination with binimetinib | Approximately 36 months
  Measure TTR